CLINICAL TRIAL: NCT02399280
Title: Effect of High Caloric Intake at Lunch Against Dinner on Weight Loss of Overweight and Obese Women Attending a Weight Loss Program, a Randomized Clinical Trial
Brief Title: Effect of High Caloric Intake at Lunch Against Dinner on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-106
Record Dates: First submitted 2015-03-22; First posted 2015-03-26 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Overweight
Keywords: Meal pattern; weight loss; high caloric intake; Dinner; Lunch
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Lunch; Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lunch (Experimental): Lunch as main meal(LM)+ Diet
  Interventions: Behavioral: Lunch as main meal(LM)+ Diet
- Dinner (Experimental): Dinner as main meal(DM)+ Diet
  Interventions: Behavioral: Dinner as main meal(DM)+ Diet

INTERVENTIONS:
Behavioral: Lunch as main meal(LM)+ Diet — Subjects are asked to have high caloric intake at lunch and low caloric intake at dinner, while they are on a multidisciplinary weight loss plan for 12 weeks.
  Arms: Lunch
Behavioral: Dinner as main meal(DM)+ Diet — Subjects are asked to have high caloric intake at dinner and low caloric intake at lunch, while they are on a multidisciplinary weight loss plan for 12 weeks.
  Arms: Dinner

SUMMARY:
The purpose of the present study is to evaluate the effect of consuming higher caloric intake at lunch in contrast to dinner on weight loss of obese and overweight female adults when they are in a multidisciplinary weight loss plan .

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks

SECONDARY OUTCOMES:
waist circumference | 12 weeks
Fasting plasma glucose level | 12 weeks
Lipid profiles | 12 weeks
Insulin resistance(HOMA) | 12 weeks
Body mass index | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Farshchi, MD, PhD, Study Chair — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ameneh Madjd, Dr., Principal Investigator — NovinDiet Clinic, School of Life Sciences, The University of Nottingham; Ian A Macdonald, Prof., Principal Investigator — School of Life Sciences, The University of Nottingham; Moira A Taylor, PhD, Principal Investigator — School of Life Sciences, The University of Nottingham; Reza Malekzadeh, Prof., Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences; Alireza Delavari, MD, Principal Investigator — Digestive Disease Research Institute, Tehran University of Medical Sciences
Locations (1):
- NovinDiet Clinic, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Madjd A, Taylor MA, Delavari A, Malekzadeh R, Macdonald IA, Farshchi HR. Beneficial effect of high energy intake at lunch rather than dinner on weight loss in healthy obese women in a weight-loss program: a randomized clinical trial. Am J Clin Nutr. 2016 Oct;104(4):982-989. doi: 10.3945/ajcn.116.134163. Epub 2016 Aug 31. PMID 27581472